CLINICAL TRIAL: NCT01118949
Title: An Open-Label Pilot Study to Assess the Safety of Oral Lacosamide as Adjunctive Therapy for Uncontrolled Primary Generalized Tonic-Clonic Seizures in Subjects With Idiopathic Generalized Epilepsy
Brief Title: Open-Label Study to Assess Lacosamide Safety as Add-on Therapy for Primary Generalized Tonic-Clonic Seizures in Subjects With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0961; 2014-004379-22 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-03

CONDITIONS: Epilepsy
Keywords: Primary Generalized Tonic-Clonic (PGTC) Seizures; Absence Seizures; Myoclonic Seizures; Idiopathic Generalized Epilepsy (IGE)
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsy, Idiopathic Generalized | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lacosamide (Experimental)
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide is supplied as 50 mg, 100 mg, 150 mg, and 200 mg tablets. Subjects will begin a Dose-Titration Phase of Lacosamide at 100 mg/day (50 mg bid, approx. 12 hours apart, once in the morning and once in the evening) for 1 week. Three (3) weekly increases will follow until the subject reaches a dosage of 200 mg/day, 300 mg/day, or 400 mg/day, as deemed clinically appropriate. The final titration will be followed by a 6-week Maintenance Phase. Subjects who complete the Maintenance Phase have the opportunity to enroll in an open-label extension study; those who do not enroll will begin a 3-week End-of-Study Phase when Lacosamide will be tapered off gradually at a recommended rate of 200 mg/day/week.
  Other Names: Vimpat®

SUMMARY:
The purpose is to assess the safety of Lacosamide in subjects with uncontrolled Primary Generalized Tonic-Clonic (PGTC) seizures with Idiopathic Generalized Epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of uncontrolled epilepsy with primary generalized tonic-clonic (PGTC) seizures and idiopathic generalized epilepsy. Diagnosis should have been established by an electroencephalogram (EEG) with generalized spike-wave discharges within 5 years of the screening visit
* Subject has ≥1 PGTC seizure within the 12 weeks prior to the screening visit
* Subject has a stable dose regimen of 1 to 3 marketed antiepileptic drug(s) (AEDs) with or without additional concurrent stable Vagus Nerve Stimulation (VNS). The VNS must have been in place for at least 6 months prior to study entry with constant settings for at least 28 days prior to the screening visit and during the Baseline Phase. Benzodiazepines will be counted as an AED

Exclusion Criteria:

* Subject has a history of partial-onset seizures or EEG findings consistent with partial onset seizures
* Subject has a history of status epilepticus within the 5-year Period prior to Visit 1
* Subject has a current or previous diagnosis of pseudoseizures, conversion disorders, or other non-epileptic ictal events
* Subject has any medical or psychiatric condition
* Subject has any history of alcohol or drug abuse
* Subject is currently taking felbamate
* Subject has ever taken vigabatrin and has no visual fields examination report available or if results of the examination are abnormal
* Subject is on a ketogenic diet
* Subject has a known sodium channelopathy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (25):
- United States (25):
  - Alabaster, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - San Francisco, California
  - Aurora, Colorado
  - Atlanta, Georgia
  - Rome, Georgia
  - Boise, Idaho
  - Fort Wayne, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Scarborough, Maine
  - Bethesda, Maryland
  - Chesterfield, Missouri
  - New York, New York
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Renton, Washington
  - Madison, Wisconsin

REFERENCES:
- [Result] Wechsler RT, Yates SL, Messenheimer J, Leroy R, Beller C, Doty P. Lacosamide for uncontrolled primary generalized tonic-clonic seizures: An open-label pilot study with 59-week extension. Epilepsy Res. 2017 Feb;130:13-20. doi: 10.1016/j.eplepsyres.2016.12.015. Epub 2016 Dec 29. PMID 28086164
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety Set (SS) includes all enrolled subjects who took at least 1 dose of Lacosamide (LCM).
Pre-assignment Details: Participant Flow and Baseline Characteristics refer to the Safety Set (SS).
Period: Overall Study
Arm/Group | Lacosamide
Started | 49
Completed | 40
Not Completed | 9
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lacosamide
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 46
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 13
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 168.08 (9.32)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 77.90 (19.80)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Seizure Days With Absence Seizures From the Baseline Phase to the Maintenance Phase
Description: During the study subjects kept a diary to record daily seizure activity from Visit 1 until the end of study participation. The following information has been recorded:
  * Seizure type
  * Seizure frequency
  A negative value in change of seizure days with absence seizures shows a decrease in seizure days with absence seizures.
Time Frame: From Baseline Phase (Weeks 0 to 4) to Maintenance Phase (Weeks 8 to 13)
Population: Of the 49 subjects in the Safety Set (SS), 44 are included in this analysis. Data not available for 5 subjects.
Measure: Mean (Standard Deviation); unit: number of seizure days
Arm/Group | Lacosamide
Number analyzed (Participants) | 44
number of seizure days | -0.37 (4.8)

2. Primary Outcome: Change in the Number of Seizure Days With Myoclonic Seizures From the Baseline Phase to the Maintenance Phase
Description: During the study subjects kept a diary to record daily seizure activity from Visit 1 until the end of study participation. The following information has been recorded:
  * Seizure type
  * Seizure frequency
  A negative value in change of seizure days with myoclonic seizures shows a decrease in seizure days with myoclonic seizures.
Time Frame: From Baseline Phase (Weeks 0 to 4) to Maintenance Phase (Weeks 8 to 13)
Population: Of the 49 subjects in the Safety Set (SS), 44 are included in this analysis. Data not available for 5 subjects.
Measure: Mean (Standard Deviation); unit: number of seizure days
Arm/Group | Lacosamide
Number analyzed (Participants) | 44
number of seizure days | -2.19 (5.80)

3. Secondary Outcome: Changes in Count of Generalized Spike-wave Discharges on 24-hour Ambulatory Electroencephalogram (EEG) From Visit 2 (Baseline Phase) to Visit 6 (Maintenance Phase)
Description: Subjects were asked to return to the clinic on the morning of the day prior to Visit 2 and Visit 6 to begin 24-hour ambulatory EEG recordings for evaluation of spike-wave discharges. Only subjects with an evaluable EEG measurement with > 19 interpretable hours at Visit 2 and Visit 6 are included in this analysis. The general spike-wave discharges are calculated per interpretable hours.
Time Frame: From Visit 2 (Week 4) to Visit 6 (Week 8)
Population: Of the 49 subjects in the Safety Set (SS), 40 subjects are included in this analysis. Data not available for 9 subjects.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Lacosamide
Number analyzed (Participants) | 40
1/hour | -3.47 (55.85)

4. Secondary Outcome: Changes in Count of 3 Hertz (Hz) Spike-wave Discharges (During Waking Hours) on 24-hour Ambulatory Electroencephalogram (EEG) From Visit 2 (Baseline Phase) to Visit 6 (Maintenance Phase)
Description: Subjects were asked to return to the clinic on the morning of the day prior to Visit 2 and Visit 6 to begin 24-hour ambulatory EEG recordings for evaluation of spike-wave discharges. Only subjects with an evaluable EEG measurement with > 19 interpretable hours at Visit 2 and Visit 6 are included in this analysis. The 3 Hertz (Hz) spike-wave discharges are calculated per awake hours.
Time Frame: From Visit 2 (Week 4) to Visit 6 (Week 8)
Population: Of the 49 subjects in the Safety Set (SS), 40 subjects are included in this analysis. Data not available for 9 subjects.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Lacosamide
Number analyzed (Participants) | 40
1/hour | 0.13 (2.17)

5. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) During the 10-week Treatment Period
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Time Frame: From Visit 2 (Week 4) to Visit 7 (Week 13)
Population: All 49 subjects in the Safety Set (SS) are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 49
participants | 43

6. Secondary Outcome: Number of Subjects Withdrawn From the Study Due to Treatment Emergent Adverse Events (TEAEs) During the 10-week Treatment Period
Description: as for outcome 5
Time Frame: From Visit 2 (Week 4) to Visit 7 (Week 13)
Population: All 49 subjects in the Safety Set (SS) are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 49
participants | 5

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 16 weeks from Baseline (Week 0 - Week 4) over the 3-weeks Titration Period (Week 4 - Week 7) and the 6-weeks Maintenance Period (Week 7 - Week 13) to the Final Clinic Visit at the end of Week 16.
Description: Adverse Events refer to the Safety Set (SS). SS includes all enrolled subjects who received at least one dose of trial medication.
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 1/49
Other Adverse Events (participants affected / at risk) | 39/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=49)
Petit mal epilepsy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=49)
Diplopia (Eye disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 13 (15)
Vomiting (Gastrointestinal disorders) | 7 (9)
Fatigue (General disorders) | 6 (6)
Gait Disturbance (General disorders) | 5 (5)
Chills (General disorders) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 3 (4)
Dizziness (Nervous system disorders) | 19 (27)
Headache (Nervous system disorders) | 8 (8)
Somnolence (Nervous system disorders) | 8 (8)
Tremor (Nervous system disorders) | 6 (8)
Migraine (Nervous system disorders) | 4 (4)
Petit mal epilepsy (Nervous system disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days